CLINICAL TRIAL: NCT07116564
Title: Impact of Multimodal Analgesia and ERAS Protocol on Length of Hospital Stay After Laparoscopic Gynecological Surgeries: A Randomized Control Trial
Brief Title: Impact of ERAS Protocol on Length of Hospital Stay After Laparoscopic Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ali Sarfraz Siddiqui, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-11268-35403
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: ERAS
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator)
  Interventions: Drug: Control
- Group E (Experimental)
  Interventions: Drug: Enhanced Recovery After Surgery

INTERVENTIONS:
Drug: Enhanced Recovery After Surgery — Preoperatively ERAS protocol includes, No solid food for 6 hours before procedure; 800 ml (fantomalt powder) Carbohydrate drink 8 hours before surgery; 400 ml (fantomalt powder) 2 hours before surgery; Celecoxib 200g 1 hour before surgery . Intraoperatively, on induction lidocaine 1.5 mg/kg and Fentanyl 1 to 2 mcg/kg followed by IV lidocaine infusion at 1.5 mg/kg/h.
  Arms: Group E
Drug: Control — Preoperatively, NPO 6 hours before the procedure Intraoperatively, on induction Nabuphine 0.1mg/kg
  Arms: Group C

SUMMARY:
The goal of this clinical trial is to determine the length of hospital stay in patients using multimodal analgesia with or without ERAS protocol scheduled for elective laparoscopic gynecological surgeries

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, and III
* Patients scheduled for elective laparoscopic gynecological surgeries

Exclusion Criteria:

* Refusal to participate
* History of allergy or contraindication to study drugs
* Patients in which procedure converted to open surgery
* Diagnostic laparoscopic procedures
* Patients with a history of severe anxiety or depression

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 98 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From arrival in the recovery room post-surgery until 72 hours after surgery.
  Post-operative length of hospital stay, measured in hours from the patient's arrival in the recovery room until 72 hours after surgery.

SECONDARY OUTCOMES:
Postoperative pain score | 4 hours, 8 hours, 12 hours, 24 hours, 48 hours & 72 hours postoperatively
  Post operative pain score will be measures using NRS (Numerical Rating Scale). Eleven points pain scale measures from 0-10, where "0" is no pain and "10" is the worst possible pain
Amount of opioid used in patient controlled analgesia | 12 hours postoperatively.
  Total Nalbuphine consumption in 12 hours (in milligrams)
Patient satisfaction Score | 24 hours after the operation
  Patient satisfaction with the pain management regimen will be assessed using a five-point Likert scale 24 hours after surgery. The scale ranges from 1 to 5, where 1 = Very Dissatisfied, 2 = Dissatisfied, 3 = Neutral, 4 = Satisfied, and 5 = Very Satisfied. Higher scores indicate greater satisfaction.

IPD SHARING:
Plan to Share IPD: Undecided